CLINICAL TRIAL: NCT00069212
Title: Psychobiological Mechanisms of Resilience to Trauma
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030292; 03-M-0292
Record Dates: First submitted 2003-09-17; First posted 2003-09-18 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2012-09-17

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Post-Traumatic Stress Disorder; Neural Circuits; Fear; Emotional Regulation; Reward; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation

SUMMARY:
This study will evaluate brain changes and psychological characteristics of people who are resilient to trauma. It will examine and compare responses in three categories of subjects: 1) people who have been exposed to a significant traumatic event and suffer symptoms of post-traumatic stress disorder (PTSD) severe enough to interfere with their ability to function; 2) people who have been exposed to a significant traumatic event and do not suffer PTSD symptoms severe enough to interfere with their ability to function; and 3) people who have never been exposed to a significant traumatic event. Most people who are exposed to trauma recover well from the adversity. Some may even benefit from it by, for example, gaining greater self-confidence of strengthening personal relationships. Others, however, develop PTSD and may have repeated thoughts, images, and dreams of the trauma; feel upset when reminded of the traumatic event; avoid places or people that remind them of the trauma; feel detached from others; have difficulty sleeping and concentrating; or startle easily.

People in the three categories listed above may be eligible for this study. Candidates will be screened with a medical and psychiatric interview, evaluation of emotional intelligence (sensitivity to feelings of others), physical examination, electrocardiogram (EKG) and blood tests.

Participants will undergo the following additional tests and procedures:

* 24-hour urine collection and three urine drug screens over the course of the study.
* Saliva collection every 2 hours on the day of the urine collection.
* Magnetic resonance imaging (MRI) scans of the brain: Subjects will have three MRI scanning sessions to show brain structure and changes in blood flow in different regions of the brain that are responsible for emotion. MRI uses a strong magnetic field and radio waves to produce images of body tissues. During the scan, the subject lies on a table in a narrow cylinder containing a magnetic field and may wear earplugs to muffle loud sounds that occur during the scanning process. While in the scanner, the subject is shown pictures of faces, houses, or words and performs tasks that involve making decisions about the pictures Subjects are also shown pleasant, unpleasant, and neutral pictures; and they are asked to play two games of chance - one that evaluates social cooperation; the other evaluating decision-making. Heart rate, blood pressure and respiration are measured during the scans.
* Neuropsychological testing: These tests are designed to evaluate memory, learning, attention and concentration, and naming.
* Aversive conditioning: This procedure examines how the body reacts to unpleasant stimuli, such as a mildly unpleasant electrical stimulation to the wrist or a loud sound, over time. During the test, heart rate, electrodermal activity (sweat), respiration, finger pulse volume, and eyeblink responses will be measured. A small blood sample will be drawn every 5 minutes to evaluate plasma levels of various stress hormones, including cortisol, neuropeptide Y, norepinephrine, and others.
* Genetic and biological testing: Patients who agree to genetic testing will have a blood sample drawn for DNA studies to better understand the biology and pharmacology of PTSD.

DETAILED DESCRIPTION:
Since the majority of research studies in posttraumatic stress disorder (PTSD) have focused on the pathological consequences of exposure to trauma, there is a paucity of information on the psychobiology of subjects who are resilient to severe stress. The proposed study will comprehensively evaluate the neural circuits that mediate fear, reward, social cooperation, memory, and emotional regulation in traumatized men and women with and without PTSD and healthy subjects. Subject groups will include prisoners of war, active duty special operations forces, returning Iraqi veterans (approval pending), and men and women exposed to non-combat traumas including sexual and or physical abuse. Comparison groups will include men and women exposed to trauma without PTSD (resilient subjects), and healthy men and women who have never been exposed to trauma. Changes in neural circuitry associated with resilience will be evaluated using functional magnetic resonance imaging (fMRI). Relationships and interactions among the neural circuits mediating fear, reward, social cooperation, memory, and emotional regulation will be assessed and correlated with clinical, neuroendocrine, and neuropsychological findings. Identification of biological and psychosocial correlates of resilience could help predict illness vulnerability following exposure to trauma and could assist in the selection of "hardy" subjects for high-risk professions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Over 18 years of age.
* Able to give written informed consent prior to participation in this study.
* Non-Combat Veterans: Not currently on medications for PTSD or other medications that would interfere with cognitive function. Patients will not be discontinued from effective medication for purposes of the study.
* Combat Veterans: Some OIF/OEF veterans may not be medication free at the time of scanning. However, they will meet criteria for PTSD according to DSM IV and meet a severity score of greater than or equal to 50 on the CAPS.
* All subjects must be in good physical health as confirmed through the screening session (under screening protocol 01-M-0254). If subjects participated in other research studies or had blood work through their primary MD within the prior 6 months, these results will be used instead of repeating blood draws for inclusion into the study. Subjects with stable medical problems will be included.
* Resilient subjects or trauma controls will be defined as those subjects who met criteria for significant trauma according to "A" criteria for PTSD (DSM-IV) but did not develop PTSD symptoms.

EXCLUSION CRITERIA:

* Have a clinically significant or unstable medical disorder.
* Meet DSM-IV criteria for alcohol and/or substance abuse or substance dependence within 6 months prior to screening.
* Currently on fluoxetine (justification: washout from fluoxetine could take up to six weeks).
* Currently at high risk for homicide or suicide.
* A current or past history of other Axis 1 disorders such as schizophrenia, schizoaffective disorder, bipolar disorder. However, those with a comorbid history of other Axis 1 disorders such as major depression, dysthymia, or panic disorder will be included. (Justification: approximately 70% of subjects with PTSD have comorbid depression and or alcohol abuse (Breslau 2001). Restricting the sample to PTSD patients without depression would not accurately reflect the biology of this disorder).
* For WRMAC study: Have donated a Red Cross unit of blood within 60 days prior to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2003-09-16; Study Completion 2012-09-17

CONTACTS AND LOCATIONS:
Overall Officials: James J Blair, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolphs R, Tranel D, Hamann S, Young AW, Calder AJ, Phelps EA, Anderson A, Lee GP, Damasio AR. Recognition of facial emotion in nine individuals with bilateral amygdala damage. Neuropsychologia. 1999 Sep;37(10):1111-7. doi: 10.1016/s0028-3932(99)00039-1. PMID 10509833
- [Background] Affleck G, Tennen H. Construing benefits from adversity: adaptational significance and dispositional underpinnings. J Pers. 1996 Dec;64(4):899-922. doi: 10.1111/j.1467-6494.1996.tb00948.x. PMID 8956517
- [Background] Affleck G, Tennen H, Croog S, Levine S. Causal attribution, perceived benefits, and morbidity after a heart attack: an 8-year study. J Consult Clin Psychol. 1987 Feb;55(1):29-35. doi: 10.1037//0022-006x.55.1.29. No abstract available. PMID 3571655